CLINICAL TRIAL: NCT03195855
Title: The Effects of Foot and Ankle Joint Mobilisation Combined With a Home Programme of Ankle Stretches on Joint Range of Motion and Forefoot Peak Plantar Pressures in People With Diabetic Peripheral Neuropathy: a Randomized Controlled Trial
Brief Title: Foot and Ankle Mobilisation in Diabetic Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, Mr Vasileios Lepesis, Podiatry Lecturer and part-time PhD student, University of Plymouth
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FHHS-228115-VL-026
Record Dates: First submitted 2017-06-13; First posted 2017-06-22 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Diabetic Peripheral Neuropathy; Limited Joint Mobility Syndrome; Ankle Joint Range of Motion; Forefoot Peak Plantar Pressure; Foot and Ankle Mobilisations; Home Exercise Programme / Stretches
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ankle and big toe mobilisations combined with home stretches (Experimental): Intervention group (n=29):
  This group will undertake talocural and 1st MTP joint mobilisations (x1/week for 6 weeks) and a 6 week home programme of stretching exercises.
  1. Mobilisations: In our study, a traction intervention consisting of two, 2-min sets of Maitland grade II joint traction will precede 2-min sets of Maitland grade III mobilisations with one minute rest in between sets. Four sets will be performed for the ankle and two for the MTP. This protocol has been used previously (19, 43). The direction of mobilisation force will be parallel to the treatment plane and perpendicular to the treatment plane during traction (75).
  2. Home Program: There will be 3 stretches prescribed (gastrocnemius, soleus and plantar fascia). Participants will be recommended to undertake three consecutive static stretches for 20-30s with a 1 minute rest period (76). Stretches will occur in standing.
  Interventions: Other: Manual therapy / joint mobilisations
- Control group of usual care including podiatry (No Intervention): Control group (n=29):
  Usual care including regular monitoring of foot health by podiatrists as indicated by NICE (NG19) guidelines (78). A review of current clinical practice within the podiatry clinic indicates that people with moderate/intermediate risk are reviewed every 3 months. Interventions include nail care, callus debridement and foot care advice.
  In both groups, interventions delivered by podiatrists in the study period will be determined from the clinic notes.

INTERVENTIONS:
Other: Manual therapy / joint mobilisations — Manual therapy is a common form of treatment employed usually by physiotherapists, in order to help increase range of motion of a specific joint region by restoring the arthrokinematic accessory gliding and rolling movement that is associated with normal joint movement. The hypothesised mechanism of action for this is that improvements of gliding and rolling will normalise osteokinematic rotation and consequently enable the normalisation of active movements. Another possible mechanism of action of mobilisations includes increasing the extensibility of the noncontractile capsular and ligamentous tissues. The effectiveness of passive accessory gliding techniques to increase joint ROM has been widely explored in the literature; with some studies revealing an increase in ankle dorsiflexion and others no change in ankle dorsiflexion. However, the subjects taking part in these studies were people without diabetes and mostly people with ankle sprains or ankle instability.
  Other Names: Home exercise programme / stretches
  Arms: Ankle and big toe mobilisations combined with home stretches

SUMMARY:
Diabetes can affect the blood supply to the nerves in the legs. When this occurs a peripheral neuropathy can occur when the nerves carrying sensory information are affected. People with diabetic peripheral neuropathy have a high risk of foot ulceration and amputation which affects function and associated with high NHS and social care costs. People with diabetes can also have reduced movement at joints caused by increased stiffness in connective tissue. Reductions in ankle and big toe movement leads to increases in the pressure over the sole on the front part of the foot (the forefoot) when walking; this is a risk factor for ulceration.

The study will to assess whether ankle and big toe joint mobilisations and home program of stretches in people with diabetic peripheral neuropathy improves joint range of motion and reduces forefoot peak pressures.

Fifty eight people with diabetic peripheral neuropathy and a moderate risk of plantar ulceration will be recruited from a local podiatry clinic. They will be randomly assigned to an intervention (29 people) or control group (29 people). We will control for between-group differences in age using a minimization process. The intervention will consist of a 6 week program of ankle and big toe joint mobilisation by a physiotherapist and home stretches. The control group will consist of usual care including podiatry interventions.

Outcome measures will be taken at baseline, post intervention and at 3 month follow up by an assessor who does not know the group allocation. Primary outcome will be ankle range while walking with secondary outcomes including big toe joint range, forefoot pressure while walking and balance.

Changes over time between the groups will be compared statistically and the relationship between ankle range of motion and peak plantar pressure will be analysed using linear regression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type I or II diabetes with a moderate risk of foot ulceration as defined by i. Detection in less than <8/10 sites on the plantar aspect of the foot using a 10 g monofilament ii. Foot deformity defined and graded using a foot deformity score previously developed for people with diabetes (54) (Attached)
* Peripheral Neuropathy- This is defined according to NICE CG19 guidelines. Here, the ability to detect a 10g monofilament (Owen Mumford "neuropen", UK) at 5 sites per foot on the plantar aspect of the toes (1,3 and 5) and metatarsophalangeal joints (1 and 5) is tested. No feeling in less than 8 sites indicates increased risk of foot ulceration (55)
* Ankle joint stiffness: Static, non-weight bearing ankle dorsiflexion will be measured using goniometry (56). Ankle joint stiffness will be defined as 0 or less ankle dorsiflexion (14, 57) due to recent evidence that these patients are more likely to exhibit limited ankle dorsiflexion of <10 degrees during gait (58).
* Hallux joint stiffness (hallux limitus): Hallux dorsiflexion will be measured using goniometry and will be defined as <10 degrees of available dorsiflexion at the hallux during weight bearing (59, 60).
* Able to walk for 10 meters with or without using a walking aid
* Able to attend 6 sessions over a 6 week period
* Age >18 yrs

Exclusion Criteria:

* Plantar Ulceration: People with a current ulceration will be excluded from the study.
* Rheumatoid arthritis, ankle and 1st MTP osteoarthritis or Dupuytren's contractures as determined from medical notes and participants subjective response.
* Excessive distal lower limb oedema preventing mobilisation rated visually according to criteria (63). People with >+2 pitting oedema in whom it is not possible to palpate the joint line will also be excluded from the study.
* History of lower limb injury in the past three months, or leg fracture/surgery in last year
* Osteoporosis as determined by the medical notes
* Prolonged (>1 yr.) history of steroid use
* Major amputation of lower limb
* Minor foot digits amputation
* Charcot arthropathy - both stages of acute (determined by the clinical signs of unilateral swelling, elevated skin temperature, erythema and joint effusion in the foot or ankle (61)) and chronic.
* Additional neurological or oncological conditions affecting the lower limb

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2022-01-02 (Actual)

PRIMARY OUTCOMES:
Change in maximum ankle range of dorsiflexion in stance phase when both feet are in contact with the ground (double support phase). | The change of maximum dorsiflexion between immediate treatment effects (week 6) and at 3-months post intervention follow-up period (week 18).

SECONDARY OUTCOMES:
Change in maximum ankle dorsiflexion during swing phase of walking as measured by 3D motion analysis. | The following measure will be taken at across two time periods: i) immediate effects after the intervention (change between week 0-6) and ii) 3-month post intervention follow up period (change between week 0-18).
Change in total ankle range of motion during the stance phase of walking as measured by 3D motion analysis | The following measure will be taken at across two time periods: i) immediate effects after the intervention (change between week 0-6) and ii) 3-month post intervention follow up period (change between week 0-18).
Walking forefoot peak plantar pressures will be measured using an in-shoe system (F Scan UK) | The following measure will be taken at across two time periods: i) immediate effects after the intervention (change between week 0-6) and ii) 3-month post intervention follow up period (change between week 0-18).
Change in maximum static ankle dorsiflexion range | The following measure will be taken at across two time periods: i) immediate effects after the intervention (change between week 0-6) and ii) 3-month post intervention follow up period (change between week 0-18).
Change in maximum 1st MTP dorsiflexion range in quiet standing | The following measure will be taken at across two time periods: i) immediate effects after the intervention (change between week 0-6) and ii) 3-month post intervention follow up period (change between week 0-18).
Walking speed -maximal walking speed over 10 m | The following measure will be taken at across two time periods: i) immediate effects after the intervention (change between week 0-6) and ii) 3-month post intervention follow up period (change between week 0-18).
Stride length | The following measure will be taken at across two time periods: i) immediate effects after the intervention (change between week 0-6) and ii) 3-month post intervention follow up period (change between week 0-18).
Walking ability | The following measure will be taken at across two time periods: i) immediate effects after the intervention (change between week 0-6) and ii) 3-month post intervention follow up period (change between week 0-18).
  12 item walking scale
Change in postural sway | The following measure will be taken at across two time periods: i) immediate effects after the intervention (change between week 0-6) and ii) 3-month post intervention follow up period (change between week 0-18).
  Postural sway will me measured with posturography
Change in functional reach test | The following measure will be taken at across two time periods: i) immediate effects after the intervention (change between week 0-6) and ii) 3-month post intervention follow up period (change between week 0-18).
  Functional reach test will be measured using a yardstick mounted on the wall at shoulder height

OTHER OUTCOMES:
To investigate the relationship between changes in static and dynamic ankle ROM | The following measures will be taken at across two time periods: i) immediate effects after the intervention (change between week 0-6) and ii) 3-month post intervention follow up period (change between week 0-18
  Linear association between change in static ankle ROM and dynamic ankle ROM
To investigate the relationship between changes in ankle ROM and balance | The following measures will be taken at across two time periods: i) immediate effects after the intervention (change between week 0-6) and ii) 3-month post intervention follow up period (change between week 0-18)
  Linear association between change in static ankle ROM and postural sway
To investigate the compliance/adherence rates of the home exercise programme | The following measure will be taken at across two time periods: i) immediate effects after the intervention (change between week 0-6) and ii) 3-month post intervention follow up period (change between week 0-18).
  Home exercise sheets diary; this will indicate any daily stretches that are undertaken, the frequency (number per day) and total duration of stretching. An open question will encourage participants to indicate any additional comments to give insight into the thinking behind why people chose to complete or not complete the stretches.The interview schedule will be generated from the recurrent themes (such as attitudes, behaviours, motivations or views on exercise) identified from the comments the participants made whilst filling in their foot and ankle exercise diaries.

CONTACTS AND LOCATIONS:
Overall Officials: Vasileios Lepesis, Principal Investigator — Plymouth University
Locations (1):
- Livewell Southwest, Plymouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lepesis V, Paton J, Rickard A, Latour JM, Marsden J. Effects of foot and ankle mobilisations combined with home stretches in people with diabetic peripheral neuropathy: a proof-of-concept RCT. J Foot Ankle Res. 2023 Dec 6;16(1):88. doi: 10.1186/s13047-023-00690-4. PMID 38057930